CLINICAL TRIAL: NCT05025514
Title: Pharmaco-epidemiological Study of COVID 19 Vaccines in Patients Undergoing Immunotherapy for Cancer. A Retrospective Open Cohort Study.
Brief Title: Retrospective Study of COVID-19 Vaccines in Patients Undergoing Immunotherapy for Cancer.
Acronym: IVACOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: University Hospital, Montpellier (Other); Institut du Cancer de Montpellier - Val d'Aurelle (Other); Centre Hospitalier de Bagnols-sur-Cèze (Unknown); Centre Hospitalier du Bassin de Thau (Unknown); University Hospital, Toulouse (Other); Centre Hospitalier de Cahors (Unknown); Centre Hospitalier d'Auch (Unknown); Centre Hospitalier Intercommunal de Castres (Unknown); Centre Hospitalier d'Albi (Unknown); Clinique Claude Bernard, Albi (Unknown); Centre Hospitalier de Bigorre - Tarbes (Unknown); Clinique La Croix du Sud Quint-Fonsegrives (Unknown); Clinique Les Cèdres Cornebarrieu (Unknown); Centre Hospitalier Ales (Unknown); CENTRE HOSPITALIER COMMINGES PYRENEES (Unknown)
Responsible Party: Sponsor
Other Study IDs: LOCAL COVID/2021/NH-001; 2021-A01144-37 (Other: RCB ID)
Record Dates: First submitted 2021-08-25; First posted 2021-08-27 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Cancer; Immunotherapy
Keywords: Cancer; Covid-19; Vaccination; Immunotherapy
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated for cancer, vaccinated or eligible for anti-COVID vaccination.: Patients undergoing treatment with anti-PD immunotherapy, anti-PDL1 or anti-CTLA4 immunotherapy for any tumour (solid, liquid) treated in the medical oncology departments of the Occitanie area.
  who have been vaccinated or who are eligible for inoculation with one of the available anti-COVID19 vaccines.

SUMMARY:
The investigators wish to set up a pharmaco-epidemiological cohort within the Hospital Territorial Groups of the Cévennes-Gard Camargue, East-Hérault and Haute-Garonne and West Tarn on a specific population, patients undergoing immunotherapy for cancer, as currently there is no data available under "real life" conditions following anti-COVID vaccination19. The hypothesis is that patients undergoing immunotherapy will not develop more vaccine-related adverse events than those observed in the efficacy and safety validation studies of the BNT162b2 mRNA Covid-19, mRNA-1273 SARS CoV-2, Oxford/AstraZeneca and Ad26COV2.S, JMJ Vaccine or J & J COVID-19 Vaccine.

DETAILED DESCRIPTION:
The recent outbreak of Coronavirus 2019 (COVID-19) caused by a new zoonotic coronavirus SARS-Cov-2 poses a major public health threat, with at least 100,000,000 people infected worldwide by the end of January 2021 and over 2 million deaths. Given the scale of the pandemic, it has become imperative to quickly develop a vaccine and over 30 vaccine candidates have entered clinical evaluation. The first vaccine to receive marketing authorization in Europe and France was an mRNA vaccine, Comirnaty® (Bnt162b2; Pfizer/BioNtech). In a Phase III study of 43,448 participants, after a median follow-up of 2 months, the number of cases of COVID-19 was 8 in the vaccine arm vs. versus 162 in the placebo arm, respectively, with 1 versus 9 serious cases (Polack et al. 2020). Adverse events occurred in more than 50% of vaccinated participants and included local reactions as well as frequent systemic reactogenicity such as fatigue and headache. Fever occurred in about 15% of the participants who received the vaccine. The second vaccine to be licensed was also an mRNA vaccine: the Moderna COVID-19 mRNA (nucleoside modified) vaccine (mRNA-1273, Moderna). A Phase III trial involving 30,420 volunteers reported efficacy and safety comparable to the Pfizer/BioNtech vaccine. A severe form of COVID-19 occurred in 30 subjects, with one death; all 30 cases were in the placebo group. Moderate and transient reactogenicity after vaccination occurred more frequently in the mRNA-1273 group.

Serious adverse events were rare and the incidence was similar in both groups. Within the vaccination strategy implemented on a national level, the Comirnaty® vaccine (Pfizer/BioNtech) and the Moderna COVID-19 mRNA vaccine (nucleoside modified) may be used interchangeably, depending on logistical constraints.

For several weeks now, the Oxford-AstraZeneca chimpanzee adenovirus vector vaccine ChAdOx1 nCoV-19 (AZD1222) has been available in France and its efficacy and safety of use have been evaluated. Also the non-replicating viral vector (adenovirus) vaccine for CVD 19 from Janssen Laboratories (a subsidiary of Johnson & Johnson; other names: Ad26COV2.S; JMJ Vaccine or J & J COVID-19 Vaccine) was launched in France a few weeks ago. Its efficacy and safety have been validated in a phase III trial. A number of other candidate vaccines using various techniques such as mRNA, protein subunit, viral vector or inactivated vaccines are currently under investigation and will be available soon.

Cancer patients are particularly at risk of developing a severe form of COVID-19. Patients with solid tumors appear to be at a greater risk, particularly in the first year after diagnosis. Severity and mortality rates in the COVID-19 and Cancer Consortium (CCC19) registry and other cohorts range from 5% to 61% (a meta-analysis showed 26%), which is well above the general population. Although data on vaccination in cancer patients are limited, there is sufficient evidence to support anti-infective vaccination in general, even in cancer patients on immunosuppressive therapy. In its notice dated January 25th, 2021, the National Cancer Institute defined its recommendations for prioritizing cancer patients for vaccination against SARS-CoV-2. This report stresses that the data acquired from science is limited in quantity and quality concerning the emerging field of vaccination against SARS-CoV-2 and even more so in sub-populations including cancer patients. It reminds us that the challenge remains to vaccinate the entire population of patients who have or have had cancer, i.e. approximately 3.8 million people.

The level of efficacy can be expected to be generally reduced in certain cancer patient populations with intense immunosuppression, such as haematopoietic stem cell transplant recipients. However, based on extrapolation of data from other vaccines and the mechanism of action of COVID-19 (non-live) vaccines, it is conceivable that the efficacy and safety of COVID-19 vaccination could be estimated to be similar to that of non-cancer patients, although data from clinical trials are lacking. The efficacy and duration of immunity in cancer patients is still unknown and unexplored. It is therefore legitimate to propose surveillance through dedicated registries and clinical trials. Furthermore, close monitoring and follow-up of cancer patients is required after COVID-19 vaccination to assess potential adverse events and measure clinical outcomes, e.g. infection, severity and mortality from COVID-19, cancer complications etc… The investigators wish to set up a pharmaco-epidemiological cohort within the Hospital Territorial Groups of the Cévennes-Gard Camargue, East-Hérault and Haute-Garonne and West Tarn on a specific population, patients undergoing immunotherapy for cancer, as currently there is no data available under "real life" conditions following anti-COVID vaccination19. Our hypothesis is that patients undergoing immunotherapy will not develop more vaccine-related adverse events than those observed in the efficacy and safety validation studies of the BNT162b2 mRNA Covid-19, mRNA-1273 SARS CoV-2, Oxford/AstraZeneca and Ad26COV2.S, JMJ Vaccine or J & J COVID-19 Vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Patient having been vaccinated or eligible for inoculation with one of the available anti-COVID19 vaccines (except live attenuated virus) while they were or are undergoing immunotherapy with anti-PD1, anti-PDL1 or anti-CTLA4 immunotherapy whatever the tumor (solid, liquid) managed within the medical oncology services of the Occitanie region.
* Patients affiliated to or beneficiaries of a health insurance scheme.
* Patients who have received written and oral information about the study and who have no objection to participation.
* Adult patients (≥ 18 years).

Exclusion Criteria:

* Patients who have been vaccinated with a live attenuated vaccine.
* Patients with a contraindication to inclusion (including hypersensitivity to the active substance or to one of the excipients, COVID+ PCR test in the last 3 months).
* Minor patients, pregnant women, parturients, nursing mothers, persons in nursing mothers, persons in emergency situations, persons unable to persons unable to express their consent and persons under persons under court protection, subguardianship or subguardianship may not be included in this research.
* Patients in an exclusion period determined by another study.
* Patients for whom it is impossible to give clear information.
* Patients who have expressed an objection to participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of all patients with cancer requiring anti-PD, anti-PDL1 or antiCTLA4 immunotherapy for any tumour (solid, liquid) who have been vaccinated or eligible for vaccination against COVID19 (of any kind, except live, attenuated virus) and treated in the medical oncology departments of the Occitanie region.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Tolerance of immunotherapy following anti-COVID-19 vaccination | 24 hours after the vaccination
  All local adverse events (pain, rashes, bruising, lymphadenopathy) and systemic adverse events (fever, headaches, fatigue, myalgia, arthralgia, nausea, shivering, diarrhoea, allergic reaction) will be recorded.
Tolerance of immunotherapy following anti-COVID-19 vaccination | 48 hours after the vaccination
  All local adverse events (pain, rashes, bruising, lymphadenopathy) and systemic adverse events (fever, headaches, fatigue, myalgia, arthralgia, nausea, shivering, diarrhoea, allergic reaction) will be recorded.
Tolerance of immunotherapy following anti-COVID-19 vaccination | 8 days after the vaccination
  All local adverse events (pain, rashes, bruising, lymphadenopathy) and systemic adverse events (fever, headaches, fatigue, myalgia, arthralgia, nausea, shivering, diarrhoea, allergic reaction) will be recorded.
Tolerance of immunotherapy following anti-COVID-19 vaccination | 24 hours after the following vaccination
  All local adverse events (pain, rashes, bruising, lymphadenopathy) and systemic adverse events (fever, headaches, fatigue, myalgia, arthralgia, nausea, shivering, diarrhoea, allergic reaction) will be recorded.
Tolerance of immunotherapy following anti-COVID-19 vaccination | 48 hours after the following vaccination
  All local adverse events (pain, rashes, bruising, lymphadenopathy) and systemic adverse events (fever, headaches, fatigue, myalgia, arthralgia, nausea, shivering, diarrhoea, allergic reaction) will be recorded.
Tolerance of immunotherapy following anti-COVID-19 vaccination | 8 days after the following vaccination
  All local adverse events (pain, rashes, bruising, lymphadenopathy) and systemic adverse events (fever, headaches, fatigue, myalgia, arthralgia, nausea, shivering, diarrhoea, allergic reaction) will be recorded.
Tolerance of immunotherapy following anti-COVID-19 vaccination | 1 month after the following vaccination
  All local adverse events (pain, rashes, bruising, lymphadenopathy) and systemic adverse events (fever, headaches, fatigue, myalgia, arthralgia, nausea, shivering, diarrhoea, allergic reaction) will be recorded.
Tolerance of immunotherapy following anti-COVID-19 vaccination | 3 months after the following vaccination
  All local adverse events (pain, rashes, bruising, lymphadenopathy) and systemic adverse events (fever, headaches, fatigue, myalgia, arthralgia, nausea, shivering, diarrhoea, allergic reaction) will be recorded.
Tolerance of immunotherapy following anti-COVID-19 vaccination | 6 months after the following vaccination
  All local adverse events (pain, rashes, bruising, lymphadenopathy) and systemic adverse events (fever, headaches, fatigue, myalgia, arthralgia, nausea, shivering, diarrhoea, allergic reaction) will be recorded.

SECONDARY OUTCOMES:
A. Tolerance of immunotherapy after anti-COVID-19 vaccination | 24 hours after the vaccination
  Any adverse events related to the immunotherapy qualified as Grade ≥3 according to the Common Terminology Criteria for Adverse Events classification (NCI CTCAE V5.0) will be recorded.
A. Tolerance of immunotherapy after anti-COVID-19 vaccination | 48 hours after the vaccination
  Any adverse events related to the immunotherapy qualified as Grade ≥3 according to the Common Terminology Criteria for Adverse Events classification (NCI CTCAE V5.0) will be recorded.
A. Tolerance of immunotherapy after anti-COVID-19 vaccination | 8 days after the vaccination
  Any adverse events related to the immunotherapy qualified as Grade ≥3 according to the Common Terminology Criteria for Adverse Events classification (NCI CTCAE V5.0) will be recorded.
A. Tolerance of immunotherapy after anti-COVID-19 vaccination | 24 hours after the following vaccination
  Any adverse events related to the immunotherapy qualified as Grade ≥3 according to the Common Terminology Criteria for Adverse Events classification (NCI CTCAE V5.0) will be recorded.
A. Tolerance of immunotherapy after anti-COVID-19 vaccination | 48 hours after the following vaccination
  Any adverse events related to the immunotherapy qualified as Grade ≥3 according to the Common Terminology Criteria for Adverse Events classification (NCI CTCAE V5.0) will be recorded.
A. Tolerance of immunotherapy after anti-COVID-19 vaccination | 1 month after the following vaccination
  Any adverse events related to the immunotherapy qualified as Grade ≥3 according to the Common Terminology Criteria for Adverse Events classification (NCI CTCAE V5.0) will be recorded.
A. Tolerance of immunotherapy after anti-COVID-19 vaccination | 3 months after the following vaccination
  Any adverse events related to the immunotherapy qualified as Grade ≥3 according to the Common Terminology Criteria for Adverse Events classification (NCI CTCAE V5.0) will be recorded.
A. Tolerance of immunotherapy after anti-COVID-19 vaccination | 6 months after the following vaccination
  Any adverse events related to the immunotherapy qualified as Grade ≥3 according to the Common Terminology Criteria for Adverse Events classification (NCI CTCAE V5.0) will be recorded.
B.Response to vaccine: dosage of anti-Spike antibodies (ELISA) | Day 0
  Quantification of anti-Spike IgG by ELISA.
B.Response to vaccine: dosage of anti-RBD antibodies (ELISA) | Day 0
  Quantification of anti-RBD IgG by ELISA.
B. Response to vaccine: Lymphocyte count by Quantiferon | Day 0
  Lymphocytes will be measured in µg/ml
B. Response to vaccine: dosage of anti-Spike antibodies (ELISA) | 1 month after the injection
  Quantification of anti-Spike IgG by ELISA.
B. Response to vaccine: dosage of anti-RBD antibodies (ELISA) | 1 month after the injection
  Quantification of anti-RBD IgG by ELISA.
B. Response to vaccine: Lymphocyte count by Quantiferon | 1 month after the injection
  Lymphocytes will be measured in µg/ml
B. Response to vaccine: dosage of anti-spike antibodies (ELISA) | 1 month after the following injection
  Quantification of anti-Spike IgG by ELISA.
B. Response to vaccine: dosage of anti-RBD antibodies (ELISA) | 1 month after the following injection
  Quantification of anti-RBD IgG by ELISA.
B. Response to vaccine: Lymphocyte count by Quantiferon | 1 month after the following injection
  Lymphocytes will be measured in µg/ml
B. Response to vaccine: dosage of anti-spike antibodies (ELISA) | 3 months after the following injection
  Quantification of anti-Spike IgG by ELISA.
B. Response to vaccine: dosage of anti-RBD antibodies (ELISA) | 3 months after the following injection
  Quantification of anti-RBD IgG by ELISA.
B. Response to vaccine: Lymphocyte count by Quantiferon | 3 months after the following injection
  Lymphocytes will be measured in µg/ml
B. Response to vaccine: dosage of anti-spike antibodies (ELISA) | 6 months after the following injection
  Quantification of anti-Spike IgG by ELISA .
B. Response to vaccine: dosage of anti-RBD antibodies (ELISA) | 6 months after the following injection
  Quantification of anti-RBD IgG by ELISA .
B. Response to vaccine: Lymphocyte count by Quantiferon | 6 months after the following injection
  Lymphocytes will be measured in µg/ml
C. Efficacy of vaccination against the incidence of COVID-19 | 1 month after vaccination
  The efficacy of vaccination against the incidence of COVID-19 will be evaluated based on the main clinical symptoms noted and a PCR test. Qualitative: YES/NO
C. Efficacy of vaccination against the incidence of COVID-19 | 3 months after vaccination
  The efficacy of vaccination against the incidence of COVID-19 will be evaluated based on the main clinical symptoms noted and a PCR test. Qualitative: YES/NO
C. Efficacy of vaccination against the incidence of COVID-19 | 6 months after vaccination
  The efficacy of vaccination against the incidence of COVID-19 will be evaluated based on the main clinical symptoms noted and a PCR test. Qualitative: YES/NO
D. Constitution of a biobank | Up to 6 months after vaccination
  Unused sample aliquots (tube bottoms) at the end of the tests will be kept; constitution of a serum library and an immune bank. Samples will be stored at -80°C (plasma) and -196°C (Peripheral Blood Mononuclear Cells) at the Biological Resource Centre at Nîmes University Hospital.

OTHER OUTCOMES:
Sex of patients | Day 0
  Male/Female
Age of patients | Day 0
  In years
Weight of patients | Day 0
  In kilograms
Height of patients | Day 0
  In centimeters
Patients' WHO status | Day 0
  The clinical status on the WHO COVID-19 ordinal scale. The WHO ordinal scale ranges from 0 to 8 in which 0 = no COVID-19 infection and 8 = death
Type of cancer and its location | Day 0
  The type of cancer and its location will be recorded
Treatment type | Day 0
  The type of treatment will be recorded
Therapeutic line | Day 0
  The therapeutic line will be noted
Other vaccinations | Day 0
  All vaccinations received other than anti-COVID-19 in the previous 6 months will be recorded.
Lymphocyte count | Day 0
  A lymphocyte count will be made at the time of vaccination and measured as the number of cells/μL
COVID-19 serology test | Day 0
  A COVID-19 serology test will be made and COVID-19-specific antibodies will be measured in μg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Nadine HOUEDE, Professeur, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (13):
- France (13):
  - Clinique Claude Bernard, Albi
  - Centre Hospitalier d'Albi, Albi
  - Centre Hospitalier d'Alès, Alès
  - CH d'Auch, Auch
  - CH de Bagnols sur Cèze, Bagnols-sur-Cèze
  - CH de Cahors, Cahors
  - Clinique des Cèdres - Capio, Cornebarrieu
  - Institut de Cancer de Montpellier, Montpellier
  - Clinique La Croix du Sud, Quint-Fonsegrives
  - Centre Hospitalier COMMINGES PYRENEES, Saint-Gaudens
  - Centre Hospitalier du bassin de Thau, Sète
  - CH de Bigorre, Tarbes
  - Centre Hospitalier de Toulouse, Toulouse

REFERENCES:
- [Background] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Background] Knoll MD, Wonodi C. Oxford-AstraZeneca COVID-19 vaccine efficacy. Lancet. 2021 Jan 9;397(10269):72-74. doi: 10.1016/S0140-6736(20)32623-4. Epub 2020 Dec 8. No abstract available. PMID 33306990
- [Background] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989
- [Background] Sadoff J, Gray G, Vandebosch A, Cardenas V, Shukarev G, Grinsztejn B, Goepfert PA, Truyers C, Fennema H, Spiessens B, Offergeld K, Scheper G, Taylor KL, Robb ML, Treanor J, Barouch DH, Stoddard J, Ryser MF, Marovich MA, Neuzil KM, Corey L, Cauwenberghs N, Tanner T, Hardt K, Ruiz-Guinazu J, Le Gars M, Schuitemaker H, Van Hoof J, Struyf F, Douoguih M; ENSEMBLE Study Group. Safety and Efficacy of Single-Dose Ad26.COV2.S Vaccine against Covid-19. N Engl J Med. 2021 Jun 10;384(23):2187-2201. doi: 10.1056/NEJMoa2101544. Epub 2021 Apr 21. PMID 33882225
- [Background] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Background] Anderson EJ, Rouphael NG, Widge AT, Jackson LA, Roberts PC, Makhene M, Chappell JD, Denison MR, Stevens LJ, Pruijssers AJ, McDermott AB, Flach B, Lin BC, Doria-Rose NA, O'Dell S, Schmidt SD, Corbett KS, Swanson PA 2nd, Padilla M, Neuzil KM, Bennett H, Leav B, Makowski M, Albert J, Cross K, Edara VV, Floyd K, Suthar MS, Martinez DR, Baric R, Buchanan W, Luke CJ, Phadke VK, Rostad CA, Ledgerwood JE, Graham BS, Beigel JH; mRNA-1273 Study Group. Safety and Immunogenicity of SARS-CoV-2 mRNA-1273 Vaccine in Older Adults. N Engl J Med. 2020 Dec 17;383(25):2427-2438. doi: 10.1056/NEJMoa2028436. Epub 2020 Sep 29. PMID 32991794